CLINICAL TRIAL: NCT05659758
Title: Is Effective Preoxygenation in Elderly Patients Related to Position?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Namik ozcan, Associate Professor of Anesthesiology and Reanimation, Principle Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E1-22-2775
Record Dates: First submitted 2022-12-11; First posted 2022-12-21 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Anesthesia Intubation Complication
Keywords: preoxygenation, elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Other): patients will be preoxygenated in supine position
  Interventions: Procedure: Head up positioning during preoxygenation
- 20 degree (Experimental): patients will be preoxygenated in 20 degrees head up position
  Interventions: Procedure: Head up positioning during preoxygenation
- 30 degree (Experimental): patients will be preoxygenated in 30 degrees head up position
  Interventions: Procedure: Head up positioning during preoxygenation

INTERVENTIONS:
Procedure: Head up positioning during preoxygenation — patients will be preoxygenated in head up position

SUMMARY:
The purpose of this study is to investigate the effect of the head-up position of 20 and 30 degrees on the ETO2 reaching time of 85% and the desaturation time of 92% after intubation in elderly patients compared to the supine position.

DETAILED DESCRIPTION:
Patients will be randomized into 3 groups. The patients will lay in the supine position, in the control group and 20 and 30 degrees head up position in other two groups. Each patient will be preoxygenated with well fitting anaesthesia face mask with FiO2 of 100% at least 6L of flow until the ETO2 reaches concentration of 85%. The angle (20 or 30 degrees) formed by the patients' bodies (hips and feet parallel to the ground, lifting the back from the ground plane) with the ground will be measured with a spirit level, angle meter, and confirmed with a smartphone application. The time to reach ETO2 85% by starting preoxygenation in patients will be measured and recorded with a stopwatch. When the target is reached, anesthesia induction will be performed and the patients will be intubated. After the start of the intubation attempt, the stopwatch will be started again, after intubation, the patient will be ventilated with a balloon once and the location of the tube will be confirmed, the circuit will be separated and SpO2 will be expected to go down to the level of 92 % and recorded during this time.

ELIGIBILITY:
Inclusion Criteria:

* Age above 65 years
* ASA 1-2

Exclusion Criteria:

* heart failure
* uncooperative
* patients refusing well fitting face mask before reaching EtO2 85%
* chronic lung disease
* anemia (hb<8gr/dl)
* BMI>40
* neurological sequela

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 156 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Time ETO2 85% | Time between placement of face mask and end tidal oxygen concentration reaches 85 %
  Time to reach ETO2 85 %

SECONDARY OUTCOMES:
Desaturation time | Time between initiation laryngoscopy for endotracheal intubation and peripheral oxygen saturation reaches 92 % measured by pulseoxymeter
  Time to reach the Spo2 of 92 % after intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)